CLINICAL TRIAL: NCT02453737
Title: A Phase II Study of Accelerated 3 Fraction Photon and Proton Partial Breast External Beam Radiotherapy and Partial Breast Brachytherapy for Early Invasive and Noninvasive Breast Cancer
Brief Title: A Study of Accelerated 3 Fraction Photon,Proton or Brachytherapy for Early Invasive and Noninvasive Breast Ca
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-002566; NCI-2017-02363 (Other: CTRP (Clinical Trials Reporting Program)); MC1532 (Other: Mayo Clinic); NCT03391388 (obsolete NCT alias)
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Results first posted 2023-08-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Proton; Brachytherapy; Partial Breast Irradiation; 3D Conformal Photon
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy, Conformal; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Catheter-based brachytherapy APBI (Other): 7 Gy x 3 fractions
  Interventions: Radiation: Brachytherapy APBI
- 3D-CRT APBI (Other): 7.3 Gy x 3 fractions
  Interventions: Radiation: 3D-CRT (photon) APBI
- Proton APBI (Other): 7.3 Gy x 3 fractions
  Interventions: Radiation: Proton APBI

INTERVENTIONS:
Radiation: Brachytherapy APBI
  Arms: Catheter-based brachytherapy APBI
Radiation: 3D-CRT (photon) APBI
  Arms: 3D-CRT APBI
Radiation: Proton APBI
  Arms: Proton APBI

SUMMARY:
This is an open label phase II study to determine the safety and efficacy of a novel 3 fraction daily dosing regimen for accelerated partial breast irradiation (APBI) for early invasive and noninvasive breast cancer. The three techniques utilized are recognized as standard options for the delivery of APBI, and there is no evidence that either technique is superior or inferior to any other. The APBI technique utilized will be at the physician's discretion and will be based on technical considerations, availability at the treating radiation facility, insurance coverage, as well as patient preference.

ELIGIBILITY:
Inclusion Criteria:

* Female Age ≥ 50 years at diagnosis
* Grade 1-3 invasive ductal, mucinous, tubular, colloidal, or pure ductal carcinoma in situ (DCIS) measuring ≤ 2cm (clinical stage T1).
* Estrogen Receptor (ER)+ (ER- DCIS meeting other eligibility criteria are eligible)
* Unicentric: Patients with microscopic multifocality are eligible as long as the total pathologic tumor size is <2cm.
* Surgical treatment of the breast must have been lumpectomy.
* The final margins of the resected specimen must be histologically free of tumor.
* Pathologically node negative Note: For patients with T1a, T1b, T1c invasive breast cancer (except T1mi), an axillary staging procedure should be performed (either sentinel lymph node biopsy alone or axillary dissection and the axillary node must be pathologically negative). Patients with N0 (i+) tumors on sentinel lymph node mapping or dissection (i.e., if the tumor deposit is 0.2mm or less as determined by immunohistochemistry or hematoxylin and eosin staining) will also be eligible.
* ECOG Performance Status of 0 or 1
* Negative pregnancy test done ≤7 days prior to registration, for women of childbearing potential only.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Ability to elect radiotherapy care in conjunction with their physician
* Able and willing to provide written informed consent
* Willingness to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).
* Willing to provide tissue and blood samples for correlative research purposes
* Willing to sign consent onto the Mayo Clinic Radiotherapy Patient Outcomes Registry and Biobanking study, IRB number 15-000136

Exclusion Criteria:

* Any of the following because this study involves therapy that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception
* Neoadjuvant chemotherapy
* Prior history of ipsilateral breast cancer
* Prior radiation therapy to the ipsilateral breast or thorax
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Active collagen-vascular disease that, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.
* Paget's disease of the breast
* Proven multicentric carcinoma (DCIS or invasive) in more than one quadrant or separated by 4 or more centimeters or diffuse (>1 quadrant) suspicious calcifications
* Histologic evidence of angiolympatic invasion (ALI). Note: Cases termed focally suspicious for ALI but where no definitive ALI is found are eligible.
* Surgical margins that cannot be microscopically assessed or that are positive
* Pathologic tumor >2cm in size
* Metastatic disease
* Patients for whom the delivery of APBI is not feasible or any of the dosimetric treatment criteria in section 9.7 have not been met.
* BRCA 1/2 mutation Note: Patients are not required to undergo BRCA1 and BRCA2 or other genetic mutation tests in order to enroll on the study. However, in the event a patient is tested and is found to be a mutation carrier, she would be excluded from the study.
* Breast implants (patients who have had implants removed are eligible).
* Extensive intraductal component
* Active connective tissue disease
* Reduction mammoplasty if 3DCRT or proton APBI are planned
* Last surgery >10 weeks from enrollment

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2022-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mutter, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 170 Patients were registered, but 4 patients weren't assigned to a treatment.
Groups:
- Catheter-based Brachytherapy APBI: 7 Gy x 3 fractions
  >
  > Brachytherapy APBI
- 3D-CRT APBI: 7.3 Gy x 3 fractions
  * D-CRT (photon) APBI
- Proton APBI: 7.3 Gy x 3 fractions >
  > Proton APBI
Period: Overall Study
Arm/Group | Catheter-based Brachytherapy APBI | 3D-CRT APBI | Proton APBI
Started | 56 | 58 | 52
Completed | 56 | 56 | 49
Not Completed | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Population: 4 Patients were not assigned treatment
Groups:
- Catheter-based Brachytherapy APBI: 7 Gy x 3 fractions>
  > Brachytherapy APBI
- 3D-CRT APBI: 7.3 Gy x 3 fractions>
  > 3D-CRT (photon) APBI
- Proton APBI: 7.3 Gy x 3 fractions>
  > Proton APBI
- Total: Total of all reporting groups
Arm/Group | Catheter-based Brachytherapy APBI | 3D-CRT APBI | Proton APBI | Total
Number analyzed (Participants) | 56 | 58 | 52 | 166
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.0 [60.7 to 70.3] | 66.2 [58.7 to 74.5] | 67.4 [61.9 to 76.0] | 66.8 [60.6 to 71.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 58 | 52 | 166
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 50 | 52 | 48 | 150
  Unknown or Not Reported | 6 | 4 | 4 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 54 | 52 | 50 | 156
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 1 | 6
Laterality [Count of Participants; unit: Participants]
  Right | 27 | 26 | 30 | 83
  Left | 29 | 32 | 22 | 83
Histology (grouped) [Count of Participants; unit: Participants]
  DCIS | 11 | 16 | 10 | 37
  Invasive carcinoma | 45 | 42 | 42 | 129
Histology [Count of Participants; unit: Participants]
  IDC | 44 | 36 | 35 | 115
  DCIS | 11 | 16 | 10 | 37
  Mucinous | 1 | 0 | 2 | 3
  ILC | 0 | 1 | 2 | 3
  Invasive mammary carcinoma | 0 | 5 | 3 | 8
Grade [Count of Participants; unit: Participants] — Grade I: cancer is slower-growing and less likely to spread. Grade II: cancer is growing faster than a grade 1 cancer but slower than a grade 3 cancer.
  Grade III: cancer is faster-growing that's more likely to spread.
  Participants
    Grade I | 25 | 17 | 18 | 60
    Grade II | 25 | 30 | 29 | 84
    Grade III | 4 | 7 | 5 | 16
    Unknown | 1 | 4 | 0 | 5
T-stage [Count of Participants; unit: Participants] — T1a-b: tumor that is larger than 1 mm but 10 mm or smaller. T1c: tumor that is larger than 10 mm but 20 mm or smaller. T2: tumor is larger than 20 mm but not larger than 50 mm. Tis: The cancer is confined within the ducts of the breast tissue and has not spread into the surrounding tissue of the breast.
  Participants
    T0 | 1 | 1 | 0 | 2
    Tis | 10 | 14 | 10 | 34
    T1 | 0 | 1 | 0 | 1
    T1a | 8 | 6 | 6 | 20
    T1b | 26 | 12 | 6 | 44
    T1c | 10 | 21 | 27 | 58
    T2 | 1 | 2 | 3 | 6
ER Status [Count of Participants; unit: Participants]
  Positive | 55 | 56 | 50 | 161
  Negative | 1 | 1 | 2 | 4
Ki67 value (%) [Median (Inter-Quartile Range); unit: percentage of cells] — The Ki-67< 5 is low and Ki-67 > 30 is high
  percentage of cells | 9.2 [5.8 to 15.2] | 10.6 [8.6 to 19.6] | 13.1 [6.0 to 17.5] | 10.0 [6.0 to 17.6]

OUTCOME MEASURES:

1. Primary Outcome: Change in the Rate of Adverse Cosmesis (Defined as Fair or Poor Cosmesis) Compared to Baseline Using the Harvard Cosmetic Rating:
Description: Participants end up being rated as fair or poor cosmesis from baseline.
  Excellent: treated breast nearly identical to untreated breast Good: treated breast slightly different than untreated (minimal but identifiable effects of the treated breast) Fair: Treated breast clearly different from untreated but not seriously distorted (significant radiation effects readily observable) Poor: Treated breast seriously distorted (severe sequelae of breast tissue secondary to radiation effects)
Time Frame: Baseline, 3 years
Population: At 3 years, 131 patients were evaluated for adverse cosmesis.
Measure: Count of Participants; unit: Participants
Arm/Group | Catheter-based Brachytherapy APBI | 3D-CRT APBI | Proton APBI
Number analyzed (Participants) | 46 | 47 | 38
Participants | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: 3 patients were not assessed for AEs after baseline
Groups:
- Catheter-based Brachytherapy APBI: Brachytherapy APBI
- 3D-CRT APBI: 3D-CRT (photon) APBI
- Proton APBI: Proton APBI
Arm/Group | Catheter-based Brachytherapy APBI | 3D-CRT APBI | Proton APBI
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/58 | 1/52
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/57 | 1/50
Other Adverse Events (participants affected / at risk) | 44/56 | 42/57 | 39/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter-based Brachytherapy APBI (N=56) | 3D-CRT APBI (N=57) | Proton APBI (N=50)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter-based Brachytherapy APBI (N=56) | 3D-CRT APBI (N=57) | Proton APBI (N=50)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (5) | 6 (7) | 4 (4)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Breast infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 13 (15) | 18 (18) | 25 (28)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 30 (57) | 14 (17) | 17 (22)
ECG QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 4 (11) | 9 (11) | 3 (4)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 17 (22) | 14 (17) | 16 (19)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 16 (18) | 11 (14) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT02453737/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT02453737/ICF_001.pdf